CLINICAL TRIAL: NCT05570630
Title: VAX-MOM COVID-19: Increasing Maternal COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Cynthia Rand, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007624
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Immunization; Infection; Pregnancy Related; COVID-19
Keywords: COVID-19; Vaccination; Prenatal Care
MeSH Terms: conditions — Infections; COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAX-MOM COVID-19 Intervention (Experimental)
  Interventions: Behavioral: VAX-MOM COVID-19 Intervention
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: VAX-MOM COVID-19 Intervention — The multi-component VAX-MOM COVID-19 intervention will be comprised of: training in communication, provider prompts, standing orders, and feedback on vaccination rates.
  Arms: VAX-MOM COVID-19 Intervention
Other: Standard of Care — Standard vaccine education and processes provided to patients by obstetric practices.
  Arms: Standard of Care

SUMMARY:
COVID-19 infection during pregnancy is associated with increased risk of pre-eclampsia, preterm birth and stillbirth. Pregnant people with COVID-19 have a higher rate of ICU admission and intubation than those who are not pregnant. COVID-19 vaccine is recommended before pregnancy and during pregnancy to decrease these risks. Despite the benefits of COVID-19 vaccination, only 71% of pregnant women were vaccinated for COVID-19 as of June 2022 (most prior to pregnancy), with a much lower rate of 58% among non-Hispanic Black women. An effective intervention is needed to improve COVID vaccination rates for pregnant people overall. In this study, the investigators will perform a randomized controlled trial aimed at practice change in obstetricians' offices, with an overall goal of increasing maternal COVID-19 vaccination rates.

DETAILED DESCRIPTION:
COVID-19 infection during pregnancy is associated with increased risk of pre-eclampsia, preterm birth and stillbirth. Pregnant people with COVID-19 have a higher rate of ICU admission and intubation than those who are not pregnant. COVID-19 vaccine is recommended before pregnancy and during pregnancy to decrease these risks. Despite the benefits of COVID-19 vaccination, only 71% of pregnant women were vaccinated for COVID-19 as of June 2022 (most prior to pregnancy), with a much lower rate of 58% among non-Hispanic Black women. An effective intervention is needed to improve COVID-19 vaccination rates for pregnant people overall.

Lack of vaccination stems from a combination of patient (lack of knowledge, vaccine hesitancy), provider (suboptimal communication skills, missed opportunities), and system (e.g. lack of standing orders and patient reminders) factors. An effective intervention is needed to improve COVID-19 vaccination rates for pregnant people. To address this, the investigators plan to use a clustered RCT (randomizing practices), allocating half of the participating practice sites within each health system to the VAX-MOM COVID-19 intervention and the other half to standard of care. The multi-component VAX-MOM COVID-19 intervention will be comprised of: training in communication, provider prompts, standing orders, and feedback on vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

Patient criteria:

* Sex is female
* Pregnant
* Identified as being eligible for COVID-19 vaccine

Practice personnel criteria:

*Provider, nurse or staff currently affiliated with (employed with) the participating OB/GYN sites

Exclusion Criteria:

*None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6911 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center (URMC), Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators upon request as part of a collaboration.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Practices
Period: Overall Study
Arm/Group | VAX-MOM COVID-19 Intervention | Standard of Care
Started | 4256; 14 Practices | 2655; 11 Practices
Completed | 4256; 14 Practices | 2655; 11 Practices
Not Completed | 0; 0 Practices | 0; 0 Practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAX-MOM COVID-19 Intervention | Standard of Care | Total
Number analyzed (Participants) | 4256 | 2655 | 6911
Age, Categorical [Count of Participants; unit: Participants] — Population: Demographic data was not available for one health system
  Participants
    number analyzed (Participants) | 1736 | 1765 | 3501
    <=18 years | 43 | 39 | 82
    Between 18 and 65 years | 1693 | 1726 | 3419
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4256 | 2655 | 6911
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data was missing from one health system
  Participants
    Asian: number analyzed (Participants) | 1736 | 1765 | 3501
    Asian | 47 | 69 | 116
    Black: number analyzed (Participants) | 1736 | 1765 | 3501
    Black | 319 | 367 | 686
    Hispanic: number analyzed (Participants) | 1736 | 1765 | 3501
    Hispanic | 252 | 265 | 517
    White: number analyzed (Participants) | 1736 | 1765 | 3501
    White | 931 | 892 | 1823
    Other/Unknown: number analyzed (Participants) | 1736 | 1765 | 3501
    Other/Unknown | 187 | 172 | 359
Region of Enrollment [Number; unit: participants]
  United States | 4256 | 2655 | 6911

OUTCOME MEASURES:

1. Primary Outcome: Rate of COVID-19 Vaccination (6 Month)
Description: Average rate of COVID-19 vaccination will be compared between intervention and control arms, for vaccine eligible patients at participating OB/GYN practice sites. Vaccination status will be obtained from patient electronic health records.
Time Frame: 6 months
Population: 6 month cohort
Measure: Count of Participants; unit: Participants
Arm/Group | VAX-MOM COVID-19 Intervention | Standard of Care
Number analyzed (Participants) | 2789 | 1759
Participants | 251 | 130

2. Secondary Outcome: Rate of COVID-19 Vaccination (9 Month)
Description: as for outcome 1
Time Frame: 9 months
Population: 9 month cohort
Measure: Count of Participants; unit: Participants
Arm/Group | VAX-MOM COVID-19 Intervention | Standard of Care
Number analyzed (Participants) | 4256 | 2655
Participants | 404 | 180

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | VAX-MOM COVID-19 Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT05570630/Prot_SAP_000.pdf